CLINICAL TRIAL: NCT03263624
Title: Efficacy of Combined Fractional Carbon Dioxide Laser and Topical Tazarotene in the Treatment of Psoriatic: Nail Disease a Single-blind, Intrapatient Left-to-right Controlled Study.
Brief Title: Efficacy of Combined Fractional Carbon Dioxide Laser and Topical Tazarotene in the Treatment of Psoriatic Nail Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat Mahmoud, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ltns
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Nail Psoriasis
Keywords: psoriasis; laser; nail
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): fractional carbon dioxide laser plus tazarotene 0.1% cream
  Interventions: Device: fractional carbon dioxide laser; Drug: Tazarotene Cream 0.1%
- Group (B) (Active Comparator): Tazarotene Cream 0.1%
  Interventions: Drug: Tazarotene Cream 0.1%

INTERVENTIONS:
Device: fractional carbon dioxide laser — One hand of each patient will receive three sessions of fractional carbon dioxide laser at four- week interval.
  Arms: Group (A)
Drug: Tazarotene Cream 0.1% — tazarotene cream 0.1% once daily

SUMMARY:
Nail psoriasis has a high incidence amongst patients with psoriasis.It is estimated to affect 80% of psoriatic patients at some time during their lives and has a significant adverse influence on their quality of life.

Treatment of nail psoriasis is disappointing, as it is refractory to treatment, with conventional therapies often having little effect.

DETAILED DESCRIPTION:
The characteristic lesions affecting the nail present as 'oil drop' discoloration, splinter haemorrhages, subungual hyperkeratosis, and onycholysis in the nail bed or pitting, leuconychia, erythema of the lunula and crumbling in the nail matrix.Diagnosis is customarily made by patient history and physical examination, though it may be necessary to rule out onychomycosis as a differential diagnosis.

The nail psoriasis severity index has recently been reported as a possible reproducible, objective, and simple tool for clinical assessment of psoriatic nail disease.

The modified target nail psoriasis severity index has been proposed for target nail assessment which would give a degree of gradation for each parameter of 0 to 3 (0 = none, 1 = mild, 2 = moderate, and 3 = severe) in each quadrant.The topical therapies include topical and intralesional corticosteroids , topical vitamin D3 analogues (calcipotriol) , topical tacrolimus and tazarotene[8]. The efficacy of these topical therapies in nail disease is limited mainly by the impenetrability or low penetrability of the nail and nail matrix. In patients with nail psoriasis that is resistant to topical therapies, conventional systemic therapies (e.g., phototherapy, retinoids, cyclosporine, methotrexate) have been shown to be partially effective. More recently, biological therapies (e.g., infliximab, adalimumab, alefacept, etanercept) have proven efficacy in psoriasis and psoriatic arthritis, and some are effective in treating nail disease in patients with psoriasis .

Previous study proved successful treatment of onychodystrophy using fractional carbon dioxide laser with topical steroid. Fractional Carbon dioxide laser might be an effective therapy for nail psoriasis due to its ablative ability which produce microscopic holes that perhaps improve topical drug delivery. Moreover it was hypothesized that tissue ablation and remodelling process stimulate rejuvenation of the abnormal nail bed.The investigators hypothesized that the combination of Fractional carbon dioxide laser and topical tazarotene treatment will have a higher therapeutic effect on nail psoriasis through multiple mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Thirty patients with bilateral fingernail psoriasis will be recruited from the Dermatology Outpatient Clinic, Assiut University Hospital.
2. The diagnosis will be based upon the clinical characteristics of nail psoriasis.
3. Patients will be included after they have stopped any systemic therapy for at least 8 weeks

Exclusion Criteria:

1. pregnant or lactating woman
2. patients with history of photosensitivity.
3. Patients who discontinued or just started to receive new systemic therapy or phototherapy during the study period will be dropped from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
percentage of clinically improved patients using modified nail psoriasis severity index. | three months
  clinical assessment using modified nail psoriasis severity index.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salomon J, Szepietowski JC, Proniewicz A. Psoriatic nails: a prospective clinical study. J Cutan Med Surg. 2003 Jul-Aug;7(4):317-21. doi: 10.1007/s10227-002-0143-0. Epub 2003 Jul 28. PMID 12879333
- [Background] Sanchez-Regana M, Aldunce Soto MJ, Belinchon Romero I, Ribera Pibernat M, Lafuente-Urrez RF, Carrascosa Carrillo JM, Ferrandiz Foraster C, Puig Sanz L, Dauden Tello E, Vidal Sarro D, Ruiz-Villaverde R, Fonseca Capdevila E, Rodriguez Cerdeira MC, Alsina Gibert MM, Herrera Acosta E, Marron Moya SE; en representacion del Grupo Espanol de Psoriasis de la Academia Espanola de Dermatologia y Venereologia. Evidence-based guidelines of the spanish psoriasis group on the use of biologic therapy in patients with psoriasis in difficult-to-treat sites (nails, scalp, palms, and soles). Actas Dermosifiliogr. 2014 Dec;105(10):923-34. doi: 10.1016/j.ad.2014.02.015. Epub 2014 May 19. English, Spanish. PMID 24852726
- [Background] Grover C, Reddy BS, Uma Chaturvedi K. Diagnosis of nail psoriasis: importance of biopsy and histopathology. Br J Dermatol. 2005 Dec;153(6):1153-8. doi: 10.1111/j.1365-2133.2005.06862.x. PMID 16307651
- [Background] Rich P, Scher RK. Nail Psoriasis Severity Index: a useful tool for evaluation of nail psoriasis. J Am Acad Dermatol. 2003 Aug;49(2):206-12. doi: 10.1067/s0190-9622(03)00910-1. PMID 12894066
- [Background] Cassell SE, Bieber JD, Rich P, Tutuncu ZN, Lee SJ, Kalunian KC, Wu CW, Kavanaugh A. The modified Nail Psoriasis Severity Index: validation of an instrument to assess psoriatic nail involvement in patients with psoriatic arthritis. J Rheumatol. 2007 Jan;34(1):123-9. PMID 17216680
- [Background] Oram Y, Akkaya AD. Treatment of nail psoriasis: common concepts and new trends. Dermatol Res Pract. 2013;2013:180496. doi: 10.1155/2013/180496. Epub 2013 May 13. PMID 23762032
- [Background] Jiaravuthisan MM, Sasseville D, Vender RB, Murphy F, Muhn CY. Psoriasis of the nail: anatomy, pathology, clinical presentation, and a review of the literature on therapy. J Am Acad Dermatol. 2007 Jul;57(1):1-27. doi: 10.1016/j.jaad.2005.07.073. PMID 17572277
- [Background] Lim EH, Seo YJ, Lee JH, Im M. Onychodystrophy treated using fractional carbon dioxide laser therapy and topical steroids: new treatment options for nail dystrophy. Dermatol Surg. 2013 Dec;39(12):1931-3. doi: 10.1111/dsu.12365. Epub 2013 Oct 26. No abstract available. PMID 24164919
- [Background] Rigopoulos D, Gregoriou S, Katsambas A. Treatment of psoriatic nails with tazarotene cream 0.1% vs. clobetasol propionate 0.05% cream: a double-blind study. Acta Derm Venereol. 2007;87(2):167-8. doi: 10.2340/00015555-0195. No abstract available. PMID 17340027
- [Background] Velez NF, Jellinek NJ. Response to onychodystrophy treated using fractional carbon dioxide laser therapy and topical steroids. Dermatol Surg. 2014 Jul;40(7):801-2. doi: 10.1111/DSU.0000000000000036. No abstract available. PMID 25111355
- [Background] Fischer-Levancini C, Sanchez-Regana M, Llambi F, Collgros H, Exposito-Serrano V, Umbert-Millet P. Nail psoriasis: treatment with tazarotene 0.1% hydrophilic ointment. Actas Dermosifiliogr. 2012 Oct;103(8):725-8. doi: 10.1016/j.ad.2012.04.008. Epub 2012 Jul 19. English, Spanish. PMID 22818395
- [Background] Treewittayapoom C, Singvahanont P, Chanprapaph K, Haneke E. The effect of different pulse durations in the treatment of nail psoriasis with 595-nm pulsed dye laser: a randomized, double-blind, intrapatient left-to-right study. J Am Acad Dermatol. 2012 May;66(5):807-12. doi: 10.1016/j.jaad.2011.12.015. Epub 2012 Jan 13. PMID 22243768
- [Background] Maranda EL, Nguyen AH, Lim VM, Hafeez F, Jimenez JJ. Laser and light therapies for the treatment of nail psoriasis. J Eur Acad Dermatol Venereol. 2016 Aug;30(8):1278-84. doi: 10.1111/jdv.13678. Epub 2016 May 26. PMID 27226341